CLINICAL TRIAL: NCT02737098
Title: Implementation of Telemedicine Outreach for PTSD (TOP) in Small Rural CBOCs (QUE 15-282)
Brief Title: TOP Implementation Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-005; QUE 15-282 (Other Grant/Funding Number: VA QUERI)
Record Dates: First submitted 2016-03-21; First posted 2016-04-13 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; virtual care; implementation; telepsychiatry; telepsychology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Implementation (Active Comparator): Standard VA implementation strategies will include disseminating a clinical intervention manual, a local champion guide, care manager training materials, PTSD case-finder tool, and technical support from the facility level telehealth technician. Internal facilitation will be conducted by the designated local champion. In addition, each VAMC will receive funds to hire a full time telephone care manager.
  Interventions: Other: Standard Implementation Strategy
- Enhanced Implementation Strategy (Active Comparator): The enhanced implementation strategy will add external facilitation to the standard VA implementation strategies. External facilitation will begin with an assessment of the current workflow at the VHA Medical Center and the affiliated CBOCs using System Redesign methods. The external facilitation team will then generate a clinical workflow chart that describes the current process of care. With advice from the external facilitation team, the local champion will then incorporate the clinical process of the TOP intervention into the current clinical workflow chart, making changes to the TOP intervention and/or current clinical workflow as needed. The local champion will also meet monthly with external facilitators to troubleshoot and make refinements.
  Interventions: Other: Enhanced Implementation Strategy

INTERVENTIONS:
Other: Enhanced Implementation Strategy — The enhanced implementation strategy will add external facilitation to the standard VA implementation strategies. External facilitation will begin with an assessment of the current workflow at the VHA Medical Center and the affiliated CBOCs using System Redesign methods. The external facilitation team will then generate a clinical workflow chart that describes the current process of care. With advice from the external facilitation team, the local champion will then incorporate the clinical process of the TOP intervention into the current clinical workflow chart, making changes to the TOP intervention and/or current clinical workflow as needed. The local champion will also meet monthly with external facilitators to troubleshoot and make refinements.
  Arms: Enhanced Implementation Strategy
Other: Standard Implementation Strategy — Standard VA implementation strategies will include disseminating a clinical intervention manual, a local champion guide, care manager training materials, PTSD case-finder tool, and technical support from the facility level telehealth technician. Internal facilitation will be conducted by the designated local champion. In addition, each VAMC will receive funds to hire a full time telephone care manager.
  Arms: Standard Implementation

SUMMARY:
The Veterans Health Administration (VHA) provides care to 3.3 million Veterans living in rural areas, comprising 36% of all VHA enrollees. In 1995, VHA began expanding its system of Community Based Outpatient Clinics (CBOCs) in order to improve access for the geographically dispersed Veteran population. There are now approximately 900 CBOCs delivering a range of services to approximately 64% of VHA enrollees. While these CBOCs have dramatically improved access to first class primary care services, it has been more challenging to deliver specialty mental health care to rural Veterans. Evidence based specialty mental care practices developed for large VA Medical Centers are often not feasible to deploy in small CBOCs and thus not accessible to rural Veterans. Rural Veterans with posttraumatic stress disorder (PTSD) treated at CBOCs experience little to no improvement in their symptoms over time. A major contributor of poor PTSD outcomes is that trauma-focused evidence-based psychotherapy is not being provided to Veterans in the CBOC setting. Moreover, travel barriers prevent most rural Veterans from receiving trauma-focused evidence-based psychotherapy at large VHA Medical Centers (VAMC). Telemedicine Outreach for PTSD (TOP) is a technology-facilitated virtual care clinical intervention that is designed to enhance access to evidence based psychotherapy and pharmacotherapy. The VHA Office of Rural Health and Office of Connected Health and Telehealth Services intend to deploy the TOP intervention nationally. This project will lay the ground work for this national implementation initiative.

The goal of this implementation project is to support the national deployment of the TOP intervention and evaluate its clinical effectiveness in routine care. The specific aims are to compare the cost and effectiveness of alternative implementation strategies to promote uptake of TOP and assess impact on access and PTSD outcomes.

The project will be conducted at 6 VAMCs and affiliated CBOCs without on-site psychologists trained in trauma-focused evidence-based psychotherapy. The total anticipated sample size will be 600.

The TOP clinical intervention is delivered by a virtual care team comprising a CBOC provider, and a telephone care manager, telepsychologist and telepsychiatrist located at the VAMC. The telephone care managers will coordinates care. The telepsychologists will deliver of trauma-focused evidence-based therapy. The telepsychiatrists will provide psychiatric consultation. The standard VA implementation strategy will follow standard procedures for deploy clinical practices in the VA include disseminating support materials, providing technical assistance and transfer funds to hire clinical personnel. The enhanced implementation strategy will add external facilitation to the standard VA implementation strategies. External facilitation will begin with an assessment of the current workflow at the VHA Medical Center and the affiliated CBOCs. The external facilitation team will then generate a clinical workflow chart that describes the current process of care. With advice from the external facilitation team, local staff will then incorporate the clinical process of the TOP intervention into the current clinical workflow chart.

The project will compare the standard VA implementation strategy to the enhanced implementation strategy. All VAMCs will receive the enhanced implementation strategy if they need it, but the time period during which they will receive the enhanced implementation strategy will be randomized. This will allow us to determine whether more patients are reached by the TOP intervention during standard implementation compared to enhanced implementation. This design will also allow us to document improvements in perceived access and PTSD outcomes for patients at sites that successfully implement the TOP intervention. Data will be collected from patient survey and chart review for all patients sampled for the evaluation. Participating patients will complete a baseline survey and 3 follow-up surveys. The reach implementation outcome measure will be specified as the proportion of sampled patients who received the TOP intervention. PTSD outcomes will be specified as a continuous change in patient self-reported symptom severity between baseline and follow-up. Perceived access will be measured using items specifically developed for the project. Provider adoption will be assessed with qualitative interviews of all CBOC clinicians treating a sampled patient as well as members of the TOP intervention team. Costs - The investigators will measure the cost of both implementation strategies both prospectively and retrospectively. The investigators will collect data on implementation activities during both the standard VA and enhanced implementation strategies.

DETAILED DESCRIPTION:
Background

The Veterans Health Administration (VHA) provides care to 3.3 million Veterans living in rural areas, comprising 36% of all VHA enrollees. In 1995, VHA began expanding its system of Community Based Outpatient Clinics (CBOCs) in order to improve access for the geographically dispersed Veteran population. There are now approximately 900 CBOCs delivering a range of services to approximately 64% of VHA enrollees. While these CBOCs have dramatically improved access to first class primary care services, it has been more challenging to deliver specialty mental health care to rural Veterans. Evidence based specialty mental care practices developed for large VA Medical Centers are often not feasible to deploy in small CBOCs and thus not accessible to rural Veterans. Rural Veterans with posttraumatic stress disorder (PTSD) treated at CBOCs experience little to no improvement in their symptoms over time. A major contributor of poor PTSD outcomes is that trauma-focused evidence-based psychotherapy is not being provided to Veterans in the CBOC setting. Moreover, travel barriers prevent most rural Veterans from receiving trauma-focused evidence-based psychotherapy at large VHA Medical Centers (VAMC). Telemedicine Outreach for PTSD (TOP) is a technology-facilitated virtual care clinical intervention that is designed to enhance access to evidence based psychotherapy and pharmacotherapy. The VHA Office of Rural Health and Office of Connected Health and Telehealth Services intend to deploy the TOP intervention nationally. This project will lay the ground work for this national implementation initiative.

Specific Aims

Impact Goal - The goal of this proposed Type II Hybrid effectiveness-implementation project is to support the national deployment of the TOP intervention and evaluate its clinical effectiveness in routine care.

To achieve this goal, the following three specific aims will be conducted.

SPECIFIC AIM 1 - Compare the effectiveness of a standard VA implementation strategy to an enhanced implementation strategy in promoting uptake of TOP.

Hypothesis 1 - For sites not meeting the TOP performance metric benchmark with a standard implementation strategy, those randomized to the enhanced implementation strategy will have better reach and engagement outcomes than those randomized to continued standard VA implementation. Reach is defined using two variables: 1) the likelihood of having a care manager encounter and 2) the likelihood of having an evidence based psychotherapy encounter. Engagement is defined using two variables: 1) the likelihood of having 8 care manager encounters and 2) the likelihood of having 8 evidence based psychotherapy encounters.

SPECIFIC AIM 2 - Determine if implementation of TOP in routine care improves PTSD outcomes for rural Veterans.

Hypothesis 2 -Clinical outcomes at sites with higher reach and engagement rates for care manager and evidence based psychotherapy encounters will have better PTSD outcomes and perceived access compared to sites with lower reach and engagement rates and compared to the pre-implementation period.

Hypothesis 3 - Perceived access at sites implementing TOP successfully will be improved compared to sites not implementing TOP successfully and compared to the pre-implementation period.

SPECIFIC AIM 3 - Calculate the cost of the standard and enhanced implementation strategies and estimate the population level cost effectiveness of the enhanced implementation.

Methodological Approach

Setting - The project will be conducted at 6 VAMCs. CBOCs served by these 6 VAMCs without on-site psychologists trained in trauma-focused evidence-based psychotherapy will be identified and a CBOC or combination of CBOCs with 300-400 eligible patients will be selected as the implementation site(s).

Population (for evaluation) - Using administrative data from VHA's Clinical Data Warehouse (CDW), the investigators will identify all patients at participating CBOCs whose most recent PC-PTSD screen was positive, had a VHA encounter in the past 12 months with a PTSD diagnosis, and had no specialty mental health encounters at the VAMC in the past 6 months. Eligible patients will be sampled for the evaluation from the selected CBOCs and 100 will be recruited to participate from each VAMC via opt-out letters. The total anticipated sample size will be 600. Participating patients will complete a baseline survey and 3 follow-up surveys every 9 months. Local clinicians at implementation sites will have the flexibility to decide who is eligible to receive the TOP clinical intervention, but the investigators expect there will be considerable overlap between those who are eligible for the evaluation and those considered to be eligible for the TOP intervention by local clinicians.

Telemedicine Outreach for PTSD (TOP) Intervention - TOP is delivered by a virtual care team comprising a CBOC provider, and a telephone care manager, telepsychologist and telepsychiatrist located at the VAMC. The telephone care manager activities include: education, activation, barrier assessment/resolution, medication adherence and side-effect monitoring, therapy/homework adherence monitoring and symptom monitoring. The telepsychologist activities include the delivery of trauma-focused evidence-based therapy (e.g., Cognitive Processing Therapy [CPT] or Prolonged Exposure Therapy [PE]). The telepsychiatrist activities include conducting case reviews and psychiatric consultations. The core element of the TOP intervention is a case review by the virtual care team (telephone care manager, telepsychologist and telepsychiatrist) of all patients newly enrolled in care management and all those not responding to treatment, along with documentation of the case review in the Electronic Health Record. Given the dynamic nature of technology and the high degree of variability in context across clinics, the investigators will employ methods that enable the new clinical intervention to be adapted from setting to setting and to be refined over time rather than focusing on fidelity to a manualized protocol. The telepsychiatry and telepsychology can either be delivered via interactive video to the CBOC or via clinical video telehealth to home. The Veteran and the telepsychologist can choose to use smartphone apps (CPT Coach or PE Coach) designed to augment these two trauma-focused evidence-based therapies. Care managers can also use secure messaging with patients in addition to telephone calls.

Standard VA Implementation Strategy - Standard VA implementation strategies will include disseminating a TOP clinical intervention manual, a TOP local champion guide, care manager training materials, PTSD case-finder tool (with the same inclusion/exclusion criteria used for evaluation sample), and technical support from the facility level telehealth technician. Internal facilitation will be conducted by the designated local champion. In addition, each VAMC will receive funds from the Office of Rural Health to hire a full time telephone care manager for three years devoted to managing CBOC patients with mental health disorders including PTSD.

Enhanced VA Implementation Strategy - The enhanced implementation strategy will add external facilitation to the standard VA implementation strategies. External facilitation will begin with an assessment of the current workflow at the VHA Medical Center and the affiliated CBOCs using System Redesign methods. A member of the external facilitation team will conduct site visits at each VAMC and conduct telephone interviews with CBOC staff. The member of the external facilitation team will also collaborate with the local System Redesign staff member. To assess clinical workflow, the investigators will examine the administrative structure of the clinical units, staffing patterns, scopes of practice, service mix, standard operating procedures (e.g., patient check-in, screening, referrals, coding), job descriptions and annual evaluation criteria, and use of technology including telehealth, eHealth, mHealth, and the electronic health record. For the TOP intervention, key clinical workflow elements include: 1) how patients are referred to the care managers, 2) whether care managers are located at the VISN, VAMC or CBOC and in what administrative unit they are housed, 3) what type of psychotherapy is provided at the CBOC (e.g., anger management, PTSD groups, etc.), 4) formulary restrictions and prescribing patterns, 5) how psychiatric consultations are arranged, 6) how frequently patients are seen in mental health and primary care, caseloads, and wait times, 7) appointment scheduling procedures for mental health and primary care, 8) no show rates, 9) care manager software availability, 10) use of interactive video, clinical video telehealth to home, SmartPhone apps, 10) use of psychiatric rating scales, and 11) how workload credit is distributed. The external facilitation team will then generate a clinical workflow chart that describes the current process of care. With advice from the external facilitation team, the local champion will then incorporate the clinical process of the TOP intervention (including use of technology) into the current clinical workflow chart, making changes to the TOP intervention and/or current clinical workflow as needed. The local champion will also meet monthly with external facilitators to troubleshoot and make refinements.

Project Design - A stepped wedge Sequential Multiple Assignment Randomized Trial (SMART) design will be used for this Type II Hybrid Effectiveness-Implementation project. The project will compare implementation outcomes (patient reach) of the standard VA implementation strategy to the implementation outcomes of the enhanced implementation strategy. This design will also allow us to document improvements in perceived access and PTSD outcomes for patients at sites that successfully implement the TOP intervention. The investigators will begin by collecting pre-implementation access and outcomes data from a sample of patients. In the first implementation step, all six VAMCs will conduct the standard VA implementation strategy at the selected CBOCs for nine months. At the end of the first implementation step, will collect follow-up data from the sample of patients to assess perceived access, intervention reach, and clinical effectiveness. To conduct the SMART trial design it will be necessary to specify a performance measure benchmark (i.e., tailoring variable) that will be used to determine whether the standard implementation effort is successful. The investigators will define implementation success based on the capacity of the full time care manager to enroll a prespecified number of patients. Specifically, the care manager will report the number of patients enrolled in the care management protocol to the evaluation team and implementation success will be defined as 50 enrolled patients over the 9 month period. If this performance measure benchmark is attained, the VAMC will discontinue the standard VA implementation efforts, but the investigators will continue to collect evaluation data. If the performance measure benchmark is not attained, the VAMC will be randomized to either continued standard VA implementation strategy or the enhanced implementation strategy in the next step. In the second implementation step, these VAMCs will conduct either the standard or enhanced implementation strategy at selected CBOCs for nine months. At the end of the second implementation step, the investigators will again collect follow-up data from the sample of patients to assess perceived access, intervention reach, and clinical effectiveness. If the performance measure benchmark is attained in the second step at standard or enhanced implementation sites, the VAMC will discontinue implementation efforts. If the performance measure benchmark is not attained at standard implementation sites, the VAMC will receive the enhanced implementation strategy in the next step. If the performance measure benchmark is not attained at enhanced implementation sites, the VAMC will continue to receive enhanced implementation. At the end of the third implementation step, the investigators will again collect follow-up data from the sample of patients to assess perceived access, intervention reach, and clinical effectiveness.

Outcome Measures - The evaluation of the implementation strategies will be based on the RE-AIM framework. Data will be collected from patient survey and chart review for all patients sampled for the evaluation. The reach implementation outcome measure will be specified as the proportion of sampled patients who received the core element of the TOP intervention (documentation in the electronic health record of a case review of the patient by the virtual care team). This will be assessed by chart review at three time points: 1) 9 month follow-up, 2) 20 month follow-up, and 3) 31 month follow-up. For each patient sampled, perceived access and clinical effectiveness data will be collected at four different time points: 1) pre-implementation baseline, 2) 9 month follow-up, 3) 20 month follow-up, and 4) 31 month follow-up. PTSD outcomes will be specified as a continuous change in the PCL-5 score between baseline and follow-up. Perceived access will be measured using items specifically developed for the project. Provider adoption will be assessed with qualitative interviews of all CBOC clinicians treating a sampled patient as well as members of the TOP intervention team (i.e., care manager, telepsychiatrists and telepsychologists) and the local champion. During the qualitative interviews with these CBOC and VAMC providers, the investigators will also assess barriers and facilitators to adoption, including their perceived benefits and weaknesses of the TOP intervention.

Costs - The investigators will measure the cost of both implementation strategies both prospectively and retrospectively. The investigators will collect data on implementation activities during both the standard VA and enhanced implementation strategies. These costs and activities will be assessed for the investigators' operational partners, local champions, and external facilitators, as well as personnel from the implementation sites at the VISN, VAMC, and CBOCs. The investigators will first examine the components of each implementation strategy and then identify activities for each component. These activities will include clinical workflow mapping, development of training materials, training sessions, meetings, and conference calls. The investigators will develop project logs to document these activities and time spent on each activity. The external facilitators, local champions and frontline providers on the implementation team will record the logs on a regular basis. The investigators will review meeting and conference call minutes to document time spent and attendance by the facilitation team, operational partners and clinical leaders and frontline providers. TOP intervention costs will be assessed from CDW (using provider IDs to identify TOP encounters).

Data Analysis - The stepped wedge SMART design allows us to estimate the effectiveness of the implementation strategy by comparing patient reach between groups of VAMCs randomized to standard or enhanced implementation and by comparing reach outcomes over time within the same VAMC as it is transitioned from standard implementation to enhanced implementation. Likewise, by collecting PCL-5 scores pre-baseline and again throughout each implementation step, the investigators will be able to compare access and PTSD outcomes of patients between VAMCs successfully implementing TOP to those not successfully implementing TOP and by comparing access and PTSD outcomes over time within the same VAMC as it is transitions from pre-implementation to successful implementation. This will allow us to estimate the clinical effectiveness of the TOP promising practices as implemented in routine care. Following intent to treat principals, the investigators will estimate the clinical effectiveness of TOP for the entire sample regardless of whether they were reached to generate a measure of population level effectiveness. Generalized linear models will be used to account for the clustering of patients and providers within VAMCs and CBOCs. VAMCs and CBOCs will specified as random effects and time period will be specified as a fixed effect. The reach, access and PTSD outcome regressions will be estimated using patients as the unit of analysis and data from all VAMCs will be included regardless of whether the VAMC attained the performance measure benchmark. For hypothesis 1 (reach regression), the explanatory variable will be whether the VAMC was randomized to standard VA implementation or enhanced implementation during each step. For hypothesis 2 (PTSD outcomes regression) and 3 (access regression), the explanatory variable will be whether the VAMC attained the performance measure benchmark during each time period. Using implementation and intervention cost data, the investigators will also calculate the population level cost-effectiveness of using the enhanced implementation strategy to deploy the TOP promising practice relative to the standard VA implementation strategy.

ELIGIBILITY:
Inclusion Criteria:

* PTSD Diagnosis
* Positive PTSD Screen

Exclusion Criteria:

* No specialty mental health encounters at the VAMC

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach: the proportion of sampled patients who received the core element of the TOP intervention | 33 months
  The reach implementation outcome measure will be specified as the proportion of sampled patients who received the core element of the TOP intervention (documentation in the electronic health record of a case review of the patient by the virtual care team).

SECONDARY OUTCOMES:
PTSD symptom severity | 22 months
  PTSD symptom severity will be measured using the PTSD Check List (version 5). The outcome will be the average change score on this scale (from baseline to follow-up).
Perceived travel burden: Degree to which sampled patients report that traveling interferes with getting services. | 33 months
  How much does having to travel to VA appointments interfere with getting the PTSD services you want? Would you say it? Completely interferes, Interferes a great deal, Interferes somewhat, Interferes a little bit, Does not interfere at all. The outcome will be the proportion responding that it completely interferes or interferes a great deal.
Perceived wait time: Degree to which sampled patients report that appointment wait time interferes with getting services. | 33 months
  How much does having to wait for VA appointments interfere with getting the PTSD services you want? Would you say it? Completely interferes, Interferes a great deal, Interferes somewhat, Interferes a little bit, Does not interfere at all. The outcome will be the proportion responding that it completely interferes or interferes a great deal.
Perceived trust: Degree to which sampled patients report that lack of trust in providers interferes with getting services. | 33 months
  How much does lack of trust in VA providers interfere with getting the PTSD services you want? Would you say it? Completely interferes, Interferes a great deal, Interferes somewhat, Interferes a little bit, Does not interfere at all. The outcome will be the proportion responding that it completely interferes or interferes a great deal.

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fortney, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (6):
- United States (6):
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortney JC, Rajan S, Chen JA, Campbell SB, Nolan JP, Wong E, Sayre G, Petrova V, Simons CE, Reisinger HS, Schnurr PP. A mixed-methods evaluation of why an implementation trial failed to engage veterans with posttraumatic stress disorder in trauma-focused psychotherapy. J Trauma Stress. 2023 Aug;36(4):762-771. doi: 10.1002/jts.22946. Epub 2023 Jun 27. PMID 37370238
- [Derived] Fortney JC, Rajan S, Reisinger HS, Moeckli J, Nolan JP, Wong ES, Rise P, Petrova VV, Sayre GG, Pyne JM, Grubaugh A, Simsek-Duran F, Grubbs KM, Morland LA, Felker B, Schnurr PP. Deploying a telemedicine collaborative care intervention for posttraumatic stress disorder in the U.S. Department of Veterans Affairs: A stepped wedge evaluation of an adaptive implementation strategy. Gen Hosp Psychiatry. 2022 Jul-Aug;77:109-117. doi: 10.1016/j.genhosppsych.2022.03.009. Epub 2022 Mar 26. PMID 35596963